CLINICAL TRIAL: NCT03321721
Title: Conservative Versus Suture Repair of Hand and Feet Lacerations in Children
Brief Title: Cosmetic Outcome at 4 Months in Hand and Feet Lacerations in Children: Conservative Versus Suture Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment and follow up
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Trevor Tredway, MD, Associate Professor of Pediatrics, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 26912
Record Dates: First submitted 2017-09-22; First posted 2017-10-26 (Actual); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Laceration Repair, Children; Hand Injuries; Foot Injuries
Keywords: hand; feet lacerations; children; conservative management
MeSH Terms: conditions — Hand Injuries; Foot Injuries | interventions — Sutures; Wound Healing

STUDY DESIGN:
Intervention Model Description: randomized, parallel group, comparative study
Who Masked: Outcomes Assessor
Masking Description: patients are randomized after informed consent evaluation of cosmetic outcome at 4m is blinded to researchers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- conservative (No Intervention): patient fulfilling entry criteria will be randomized to the conservative arm - no suturing
- suture (Active Comparator): patient fulfilling entry criteria will be randomized to the suture arm for repair with nylon suture material
  Interventions: Procedure: Suture for wound repair; Device: Suture for wound repair

INTERVENTIONS:
Procedure: Suture for wound repair — Repair of wound with suture
  Arms: suture
Device: Suture for wound repair — Repair of wound with suture
  Arms: suture

SUMMARY:
Hand and feet lacerations are common in children with repair often requiring conscious sedation and needle sticks for repair. Growing evidence in adults reveal that many of these small lacerations do quite well cosmetically without intervention. This randomized controlled trial will evaluated the cosmetic outcome at 4 months in two groups of children with hand or feet lacerations <2 cm comparing suturing vs conservative wound management.

DETAILED DESCRIPTION:
The purpose of this study is to compare outcomes of 2 repair methods in simple (<2cm) hand and feet lacerations in the pediatric population (2-17 yrs). Our hypothesis is that there is no statistical difference in cosmetic outcomes between suture repair and non-repair of these injuries. This study has been performed in the adult population, but has not yet been done in children. The researchers would like to be the first to show that conservative repair can be done in our pediatric population. The suture group will have their injuries repaired with non-absorbable sutures (nylon) which remain the gold standard in cosmetic repair of hands and feet. The conservative group will have identical cleaning and preparation of the wound, but the laceration will be covered with antibiotic ointment and sterile gauze without repair. Secondary outcome measure include patient satisfaction, infection rates, pain during repair, time of initial ED visit stay, and cost of supplies used in repair. Our patients will return in 10 -14 days for follow up and in 4 months for evaluation of the wound and for digital pictures to be taken of the wound. Wounds and scars will be evaluated at both 10 -14 days and 4 months by both the researchers and the parents or care givers. A satisfaction survey will be administered to the parent or guardian. At 3-4 months, digital photographs of the healing lacerations will be graded for appearance by clinicians blinded to the repair method. The initial visit will be billed to their insurance and the follow-up visits will be free.

ELIGIBILITY:
Inclusion Criteria:

* Any English-speaking child, 2 to 17 years of age that presents to the emergency department at Cardinal Glennon Children's Medical Center with a hand or foot laceration less than or equal to 2 cm is eligible for the study.

Exclusion Criteria:

* Patients will be excluded if their laceration is greater than 2 cm, have irregular borders or are, deeper than 0.5 cm.
* Wounds that are the result of a mammalian bite,
* Wounds more than minimally contaminated on visual inspection or are more than 8 hours old.
* Wounds associated with an open fracture, involve a partial amputation or involve a puncture wound.
* Wounds that involve the nailbed or a fingernail avulsion will be excluded.
* Patients with confirmed or suspected retained foreign bodies in the wound would also be excluded.
* Patients will also be excluded if hemostasis could not be attained after 15 minutes of pressure.
* Patients with complex lacerations who need plastic surgery or other sub-specialty repair will be excluded.
* Complex lacerations include: associated or suspected neurovascular, tendon, ligament, or bone injury, need for deep/multi-layer sutures will be excluded.
* Patients with known or suspected immunodeficiency, bleeding or clotting disorders, pregnancy, diabetes, renal dysfunction, or allergic reaction to local anesthesia are also excluded.
* Patients with a history of anticoagulant or chronic steroid use in the last year. Chronic steroid use is defined by use of steroids (PO, IV, IM, or topical) for more than 14 consecutive days, for more than 3 separate courses per year will be excluded.
* Foster children will also be excluded, due to complications regarding custody, consent, and follow-up issues.
* Patients with allergies to topical anesthetics solution will be excluded from the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2014-04-13 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- cardinal glennon children's hospital / Division of Emergency Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
if other facilities are performing similar studies would be happy to participate
Supporting Information: Study Protocol, ICF
Time Frame: 7/19
Access Criteria: By Appointment

RESULTS

PARTICIPANT FLOW:
Groups:
- Suture-Non Absorbable: Patient fulfilling entry criteria will be randomized to the suture arm for repair with non-absorbable (nylon) suture material
- Suture-Absorbable: Patient fulfilling entry criteria will be randomized to the suture arm for repair with absorbable) suture material
Period: Overall Study
Arm/Group | Conservative | Suture-Non Absorbable | Suture-Absorbable
Started | 4 | 10 | 12
Completed | 0 | 2 | 1
Not Completed | 4 | 8 | 11
Not completed — Lost to Follow-up | 4 | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Suture (Absorbable): Patient fulfilling entry criteria will be randomized to the absorbable suture arm for repair with absorbable suture material
- Suture (Non-Absorbable): Patient fulfilling entry criteria will be randomized to the non-absorbable suture arm for repair with non-absorbable suture material
- Total: Total of all reporting groups
Arm/Group | Conservative | Suture (Absorbable) | Suture (Non-Absorbable) | Total
Number analyzed (Participants) | 4 | 12 | 10 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Ages were not recorded on 4 participants
  years
    number analyzed (Participants) | 2 | 11 | 9 | 22
    (all) | 13 (1) | 10.3 (4.61) | 8.6 (5.65) | 9.8 (5.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 3 | 7
  Male | 4 | 8 | 7 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 12 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Cosmetic Outcome of Hand and Feet Laceration in Children : Conservative vs Suture Repair
Description: Randomized, parallel group study will compare cosmetic outcome by digital picture by blinded evaluators at 4 months post enrollment.
  The digital pictures of the laceration repairs were scored using a previously validated Visual Analogue Scale (VAS). The VAS scale is a 100-mm continuous line that is marked at the right end with "best appearance/scar"(score 100), and on the left end with "worst appearance/scar" (score 0).
Time Frame: 4 months
Population: No participants in the conservative arm/group of the study completed the study protocol. Only 1 participant in the absorbable suture arm/group of the study and 2 participants in the non-absorbable arm/group of the study completed the study protocol.
Measure: Mean (Standard Deviation); unit: Score on a scale (100-mm VAS)
Arm/Group | Conservative | Suture (Absorbable) | Suture (Non-Absorbable)
Number analyzed (Participants) | 0 | 1 | 2
Score on a scale (100-mm VAS) |  | 60 | 100 (0)

2. Secondary Outcome: Wound Healing in Hand and Feet Lacerations in Children: Conservative vs Suture Repair
Description: Wound healing by visual inspection at the first follow up visit. The wounds will be evaluated for complications that were defined a priori as follows: "wound infection" was one that required systemic antibiotics as determined by the treating attending physician; and "wound dehiscence" as a wound that required the placement of additional sutures or tissue adhesives.
  The outcome measure data is reported as the number of participants without the presence of "wound infection" or "wound dehiscence".
Time Frame: 10-14 days
Population: No participants in the conservative arm/group completed the study. 3 patients in the "absorbable arm" and 4 patients in the "non-absorbable arm" completed the first part and were present for their first follow up.1 of the 3 "absorbable arm" patients completed the entire study and 2 of the 4 "non-absorbable arm" patients completed the entire study.
Measure: Count of Participants; unit: Participants
Arm/Group | Conservative | Suture (Absorbable) | Suture (Non-Absorbable)
Number analyzed (Participants) | 0 | 3 | 4
Participants |  | 0 | 0

3. Secondary Outcome: Cosmetic Outcome of Hand and Feet Laceration in Children : Conservative vs Suture Repair
Description: Infection rate by visual inspection. The wounds will be evaluated for complications that were defined a priori as follows: "wound infection" was one that required systemic antibiotics as determined by the treating attending physician; and "wound dehiscence" as a wound that required the placement of additional sutures or tissue adhesives.
Time Frame: 10-14 days
Population: No participants in the conservative arm/group completed the study protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Conservative | Suture (Absorbable) | Suture (Non-Absorbable)
Number analyzed (Participants) | 0 | 3 | 4
Participants |  | 0 | 0

4. Secondary Outcome: Cosmetic Outcome of Hand and Feet Laceration in Children : Conservative vs Suture Repair
Description: Rate of wound dehiscence by visual inspection. The wounds will be evaluated for complications that were defined a priori as follows: "wound infection" was one that required systemic antibiotics as determined by the treating attending physician; and "wound dehiscence" as a wound that required the placement of additional sutures or tissue adhesives.
Time Frame: 10-14 days
Population: No participants in the conservative arm/group completed the study protocol
Measure: Count of Participants; unit: Participants
Groups:
- Suture (Absorbable): Patient fulfilling entry criteria will be randomized to the suture arm for repair with suture material
Arm/Group | Conservative | Suture (Absorbable) | Suture (Non-Absorbable)
Number analyzed (Participants) | 0 | 3 | 4
Participants |  | 0 | 0

ADVERSE EVENTS:
Time Frame: After patients completed their final follow up visit, they were instructed to contact the PI with any concerns about the laceration repair/wound for the time period of 1 year from date of initial repair.
Groups:
- Suture (Absorbable): Patient fulfilling entry criteria will be randomized to the suture absorbable arm for repair with absorbable suture material
- Suture (Non-Absorbable): Patient fulfilling entry criteria will be randomized to the suture non-absorbable arm for repair with non-absorbable suture material
Arm/Group | Conservative | Suture (Absorbable) | Suture (Non-Absorbable)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/4 | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT03321721/Prot_SAP_000.pdf